CLINICAL TRIAL: NCT07241520
Title: Phase III Clinical Trial to Evaluate the Efficacy and Safety of SHPL-49 Injection in the Treatment of Acute Ischemic Stroke（SAIL）- a Multicenter, Randomized, Double-blind, Parallel, Placebo-controlled Phase III Clinical Trial
Brief Title: Phase III Clinical Trial of SHPL-49 Injection in the Treatment of Acute Ischemic Stroke
Acronym: SAIL
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Hutchison Pharmaceuticals Limited (Industry)
Collaborators: Beijing Tiantan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHPL-Z003-301
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: In this double-blind study, the participant, and all relevant personnel involved with the conduct and interpretation of the study (including investigator, investigational site personnel, and the sponsor or designee's staff) will remain blinded to the identity of the Investigational Product (IP) assigned and the randomization codes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHPL-49 Injection (Experimental): 3mL/ ampoule
  Interventions: Drug: SHPL-49 Injection
- Placebo Injection (Placebo Comparator): 3mL/ ampoule
  Interventions: Drug: Placebo Injection

INTERVENTIONS:
Drug: SHPL-49 Injection — 2 ampoules of SHPL-49 Injection in 100 mL 0.9% sodium chloride will be administered as a 30-minute intravenous infusion and applied twice daily for 7 days.
  Arms: SHPL-49 Injection
Drug: Placebo Injection — 2 ampoules of Placebo Injection in 100 mL 0.9% sodium chloride will be administered as a 30-minute intravenous infusion and applied twice daily for 7days.
  Arms: Placebo Injection

SUMMARY:
This study is designed to determine the efficacy and safety of SHPL-49 intravenous infusion in acute ischemic stroke patients.

DETAILED DESCRIPTION:
The objective of this study is to determine the efficacy and safety of SHPL-49 intravenous infusion for 7 consecutive days in acute ischemic stroke patients within 8hours after onset. This study is a Phase III, multicenter, randomized, double-blind, placebo-controlled parallel design. Participants receive twice daily dosing for 7 consecutive days, or once on Day 1 and Day 8 and twice daily on Days 2 to 7, with each participant scheduled to receive 14 doses throughout the clinical trial. 1096 participants will be randomized 1:1 to SHPL-49 injection treated group and placebo group.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 years old (including upper and lower limits);
2. Clinically diagnosed as acute ischemic stroke according to the latest guidelines;
3. Patients diagnosed as acute ischemic stroke who plan to receive or have received standard intravenous thrombolysis in hospital (this research center) within 8hours of symptom onset;
4. Patients who have NIHSS score≥5 and ≤ 22 before thrombolysis;
5. Pre-stroke mRS score ≤1;
6. Patients or legally authorized representatives who are able and willing to sign informed consent.

Exclusion Criteria:

1. Complicated with intracranial hemorrhagic diseases, including hemorrhagic stroke, epidural hematoma, intracranial hematoma, ventricular hemorrhage, subarachnoid hemorrhage, etc.;
2. Severe disturbance of consciousness: patients with NIHSS 1a consciousness level item score ≥2;
3. Cerebral Computed tomography (CT) or Magnetic resonance imaging (MRI) indicated a large anterior circulation cerebral infarction (infarct area greater than 1/3 of the middle cerebral artery blood supply area);
4. Stroke with rapid improvement of symptoms before intravenous thrombolysis, or acute ischemic symptoms suspected to be caused by other causes;
5. Patients who are ready to receive or have received endovascular therapy;
6. After the onset of the disease, the drugs with neuroprotective effects which have been used: commercially available Edaravone, Edaravone and Dexborneol, Butylphthalide, Citicoline, Nimodipine, Ganglioside, Human Urinary Kallidinogenase, Cinepazide, Cattle Encephalon Glycoside and Ignotin, Fasudil, Compound Porcine Cerebroside and Ganglioside, Piracetam, Oxiracetam, Mouse Nerve Growth Factor For Injection, Cerebrolysin, Deproteinised Calf Blood Serum Injection, Deproteinised Calf Blood Extractives Injection, Ginkgolides Injection, Ginkgolides Diterpene Lactone Meglumine Injection, Ginkgo Leaf Extract and Dipyridamole Injection, Extract of Ginkgo Biloba Leaves Injection, Safflower Extract and Aceglutamide Injection, Xuesaitong Injection, Xuesaitong Soft Capsules, and injections containing any single eXtract of Chuanxiong (Chuanxiong Rhizoma), Danshen (Salviae Miltiorrhizae Radix ET Rhizoma), Hongjingtian (Rhodiolae Crenulatae Radix Et Rhizoma),or several of these Chinese herbal ingredients;
7. Patients with a history of atrial fibrillation, deep vein thrombosis of the lower extremities, pulmonary embolism or other conditions that require the use of anticoagulant drugs during administration;
8. Severe hypertension: systolic blood pressure ≥180mmHg or diastolic blood pressure ≥100mmHg after taking antihypertensive drugs before thrombolysis;
9. Severe renal insufficiency: serum creatinine >2 times upper limit of normal or creatinine clearance (CLcr) < 30mL/min (Cockcroft-Gault formula), or with other known severe renal insufficiency such as renal failure and uremia ; (Note: Cockcroft Gault formula: (1) Male: CLcr (mL/min) = [140 - age (yrs)]× body weight (kg) / [0.814 × serum creatinine (μmol/L)]; (2) female: CLcr (mL/min) = {[140 - age (years old)] by weight (kg) / [0.814 x serum creatinine (μmol/L)]} x 0.85);
10. Severe hepatic function impairment: Alanine aminotransferase (ALT) or Aspartate aminotransferase(AST) 3 times upper limit of normal, or with other known hepatic diseases such as hepatic failure, hepatic cirrhosis, portal hypertension (with esophageal varices), active hepatitis, etc.;
11. Patients with a heart function rating above Class II (according to the New York Heart Association (NYHA) heart function rating) or a history of congestive heart failure;
12. Patients with malignant tumors or undergoing anti-tumor therapy;
13. Allergic to experimental drugs or similar ingredients or materials used in imaging examinations;
14. Patients during pregnancy, lactation or planning pregnancy;
15. Patients who have a history of epilepsy or have had seizure-like symptoms at the onset of stroke, or suffer from serious mental disorders, intellectual disabilities or dementia;
16. Alcohol dependence, or drinking more than 3 units (male) or 2 units (female) of alcohol within 24 hours prior to onset (1 unit =360 mL beer or 45 mL liquor with 40% alcohol or 150 mL wine);
17. Patients have participated in other drug or non-drug clinical studies, or are participating in another clinical study within 3 months before signing informed consent form;
18. Patients have a history of severe head trauma or stroke within the past 3 months;
19. Patients are suffering from severe systemic diseases, with a life expectancy of less than 90 days;
20. Patients who are judged unsuitable for participation by the investigators in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1096 (Estimated)
Dates: Start 2025-12-08 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Modified Rankin Scale (mRS), with scores of 0-1 at Day 90 | 90±7 days
  Proportion of participants with mRS scores of 0-1 at Day 90

SECONDARY OUTCOMES:
Modified Rankin Scale (mRS), with scores at Day 90 | 90±7 days
  A shift of one or more categories to reduced functional dependence analyzed across the whole distribution of outcomes on the mRS at Day 90
Modified Rankin Scale (mRS), with scores of 0-2 at Day 90 | 90±7 days
  Proportion of participants with mRS Scores of 0-2 at Day 90
Barthel index (BI) at Day 90 | 90±7 days
  Proportion of participants with BI ≥95 at Day 90
Modified Rankin Scale (mRS), with scores of 0-1 at Day 30 | 30±3 days
  Proportion of participants with mRS Scores of 0-1 at Day 30
National Institute of Health stroke scale (NIHSS), with scores of 0-1 at Day 7 or 8 | 7 days or 8 days
  The proportion of participants with NIHSS scores of 0-1 at day 7 or 8 (at the end of the last dose)
National Institute of Health stroke scale (NIHSS) at Day 7or 8 | 7 days or 8 days
  Changes in NIHSS scores from baseline at Day 7or 8 (at the end of the last dose)
Symptomatic intracranial hemorrhage | 22-36hours after thrombolysis
  Symptomatic intracranial hemorrhage within 36 hours after thrombolysis as defined by the SITS-MOST Criteria (Safe Implementation of Thrombolysis in Stroke Monitoring Study)
Mortality | 90±7 days
  Mortality over the 90-day study period
Serious adverse events | 90±7 days
  Serious adverse events over the 90-day study period
Adverse events | 90±7 days
  Adverse events over the 90-day study period

CONTACTS AND LOCATIONS:
Overall Officials: Yongjun Wang, Master, Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Linfen Central Hospital, Linfen, Shanxi, China